CLINICAL TRIAL: NCT03139240
Title: Opioid Analgesia for MAB: A Randomized Controlled Trial
Brief Title: Opioid Analgesia for MAB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Principal Investigator, Alyssa Colwill, MD, Instructor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16845
Record Dates: First submitted 2017-04-28; First posted 2017-05-03 (Actual); Results first posted 2019-08-13 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: MAB; Pain
MeSH Terms: conditions — Pain | interventions — Oxycodone

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gestational age <7 weeks (Experimental): Women with a gestational age <7 weeks will be randomized to oxycodone 10mg oral vs placebo
  Interventions: Drug: Oxycodone 10mg oral; Other: Placebo
- Gestational age 7-10w0d (Experimental): Women with a gestational age 7-10w0d will be randomized to oxycodone 10mg oral vs placebo
  Interventions: Drug: Oxycodone 10mg oral; Other: Placebo

INTERVENTIONS:
Drug: Oxycodone 10mg oral — Oxycodone 10mg oral given for pain control in addition to standard of care medications in women undergoing medical abortion
Other: Placebo — Placebo given in addition to standard of care medications in women undergoing medical abortion

SUMMARY:
Our primary objective will be to determine if a strong opioid, oxycodone, given at a dose recommended for severe pain in addition to ibuprofen decreases maximum pain scores compared to ibuprofen and placebo in women undergoing medical abortion (MAB). Results of this study will help future providers understand whether prescribing opioids are an important adjunct for pain control in women undergoing MAB.

DETAILED DESCRIPTION:
This study will include 152 women undergoing MAB. Women will be randomized to oxycodone 10mg oral versus placebo and stratified by gestational age (<7wks, 7-10wks). The primary outcome will be maximum reported pain score measured at 6-8 hours and 24 hours after misoprostol administration.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Seeking elective medical abortion
* In good health
* Pregnancy with intrauterine gestational sac up to 10 0/7 weeks, dated by ultrasound
* Able and willing to receive text messages via phone
* Literate in English
* Able and willing to give informed consent and agree to the study terms
* Have assistance at home; no motor vehicle use while taking study medications

Exclusion Criteria:

* Lack of access to cell phone and texting capabilities
* Early pregnancy failure
* Contraindications to the study medications: Oxycodone, Ibuprofen
* Contraindications to medical abortion with Mifepristone or Misoprostol
* History of methadone or heroin use
* Used alcohol in the past 24 hours
* Used marijuana >4 times per week
* Any opioid in the past 30 days
* Using additional pain medications

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 172 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Site 1, Beaverton, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Colwill AC, Bayer LL, Bednarek P, Garg B, Jensen JT, Edelman AB. Opioid Analgesia for Medical Abortion: A Randomized Controlled Trial. Obstet Gynecol. 2019 Dec;134(6):1163-1170. doi: 10.1097/AOG.0000000000003576. PMID 31764725

RESULTS

PARTICIPANT FLOW:
Groups:
- Oxycodone: <7 Weeks of Gestation: Oxycodone 10mg oral: Oxycodone 10mg oral given for pain control in addition to standard of care medications in women undergoing medical abortion
  Women with a gestational age <7 weeks randomized to oxycodone 10mg oral
- Placebo: <7 Weeks Gestational Age; Placebo: 7-10w0d Gestational Age: Placebo: Placebo given in addition to standard of care medications in women undergoing medical abortion
  Women with a gestational age <7 weeks and women with a gestational age 7-10w0d randomized to placebo
- Oxycodone: 7-10w0d Gestational Age: Oxycodone 10mg oral: Oxycodone 10mg oral given for pain control in addition to standard of care medications in women undergoing medical abortion
  Women with a gestational age 7-10w0d randomized to oxycodone 10mg oral
Period: Overall Study
Arm/Group | Oxycodone: <7 Weeks of Gestation | Placebo: <7 Weeks Gestational Age | Oxycodone: 7-10w0d Gestational Age | Placebo: 7-10w0d Gestational Age
Started | 48 | 48 | 38 | 38
Completed | 48 | 47 | 37 | 38
Not Completed | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Oxycodone: <7 Weeks Gestational Age: Oxycodone 10mg oral: Oxycodone 10mg oral given for pain control in addition to standard of care medications in women undergoing medical abortion
  Women with a gestational age <7 weeks randomized to oxycodone 10mg oral
- Placebo: <7 Weeks Gestational Age: Placebo: Placebo given in addition to standard of care medications in women undergoing medical abortion
  Women with a gestational age <7 weeks randomized to placebo
- Oxycodone: 7-10w0d Weeks Gestational Age: Oxycodone 10mg oral: Oxycodone 10mg oral given for pain control in addition to standard of care medications in women undergoing medical abortion
  Women with a gestational age 7-10w0d randomized to oxycodone 10mg oral
- Placebo: 7-10w0d Weeks Gestational Age: Placebo: Placebo given in addition to standard of care medications in women undergoing medical abortion
  Women with a gestational age 7-10w0d randomized to placebo
- Total: Total of all reporting groups
Arm/Group | Oxycodone: <7 Weeks Gestational Age | Placebo: <7 Weeks Gestational Age | Oxycodone: 7-10w0d Weeks Gestational Age | Placebo: 7-10w0d Weeks Gestational Age | Total
Number analyzed (Participants) | 48 | 48 | 38 | 38 | 172
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 48 | 48 | 38 | 38 | 172
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 48 | 38 | 38 | 172
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Non-Hispanic | 27 | 27 | 25 | 14 | 93
  Other | 21 | 21 | 13 | 24 | 79
Region of Enrollment [Number; unit: participants]
  United States | 48 | 48 | 38 | 38 | 172

OUTCOME MEASURES:

1. Primary Outcome: Overall Maximum Self-reported Pain Score
Description: Women text responses through two surveys within 24 hours after misoprostol administration indicating their maximum self-reported pain score on an 11-point Numeric Pain Rating Scale (0 = no pain, 5 = moderate pain, and 10 = worst possible pain).
Time Frame: 24 hours after misoprostol administration
Measure: Median (Full Range); unit: units on a scale
Groups:
- Oxycodone Arm: Oxycodone 10mg oral: Oxycodone 10mg oral given for pain control in addition to standard of care medications in women undergoing medical abortion
  Women with a gestational age <7 weeks and women with a gestational age 7-10w0d randomized to oxycodone 10mg oral
- Placebo Arm: Placebo: Placebo given in addition to standard of care medications in women undergoing medical abortion
  Women with a gestational age <7 weeks and women with a gestational age 7-10w0d randomized to placebo
Arm/Group | Oxycodone Arm | Placebo Arm
Number analyzed (Participants) | 86 | 86
units on a scale | 8 [2 to 10] | 8 [1 to 10]

2. Primary Outcome: <7 Weeks of Gestation - Maximum Self-reported Pain Score
Description: as for outcome 1
Time Frame: 24 hours after misoprostol administration
Population: Participants at <7 weeks of Gestation were assessed. Participants who were "lost to follow-up" were excluded from this analysis.
Measure: Median (Full Range); unit: units on a scale
Groups:
- Oxycodone: Oxycodone 10mg oral: Oxycodone 10mg oral given for pain control in addition to standard of care medications in women undergoing medical abortion
  Women with a gestational age <7 weeks randomized to oxycodone 10mg oral
- Placebo: Placebo: Placebo given in addition to standard of care medications in women undergoing medical abortion
  Women with a gestational age <7 weeks randomized to placebo
Arm/Group | Oxycodone | Placebo
Number analyzed (Participants) | 48 | 47
units on a scale | 8 [2 to 10] | 8 [1 to 10]

3. Primary Outcome: 7-10 Weeks Gestation - Maximum Self-reported Pain Score
Description: as for outcome 1
Time Frame: 24 hours after misoprostol administration
Population: Participants at 7-10w0d of Gestation were assessed. Participants who were "lost to follow-up" were excluded from this analysis.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Oxycodone | Placebo
Number analyzed (Participants) | 37 | 38
units on a scale | 9 [2 to 10] | 8 [4 to 10]

ADVERSE EVENTS:
Time Frame: 21 days
Groups:
- Oxycodone: Oxycodone 10mg oral: Oxycodone 10mg oral given for pain control in addition to standard of care medications in women undergoing medical abortion
  Women with a gestational age <7 weeks and women with a gestational age 7-10w0d randomized to oxycodone 10mg oral
- Placebo: Placebo: Placebo given in addition to standard of care medications in women undergoing medical abortion
  Women with a gestational age <7 weeks and women with a gestational age 7-10w0d randomized to placebo
Arm/Group | Oxycodone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/86
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/86
Other Adverse Events (participants affected / at risk) | 4/86 | 2/86
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxycodone (N=86) | Placebo (N=86)
Ongoing pregnancy (Reproductive system and breast disorders) | 4 (4) | 2 (2) — Resolved with standard treatment measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-20): https://cdn.clinicaltrials.gov/large-docs/40/NCT03139240/Prot_SAP_000.pdf